CLINICAL TRIAL: NCT05819801
Title: Effect of Fasting on Patient Outcomes After Wide-Awake, Local Anesthesia-only, No Tourniquet (WALANT) Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jesse Kaplan, Assistant Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2157
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Surgery; Anesthesia, Local; Fasting
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into two groups and told whether to eat or fast prior to their procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): Patients in the fasting group will be told to avoid any food past midnight the day before their surgery and any liquids 4 hours before their scheduled surgery.
  Interventions: Other: Fasting
- Not Fasting (Experimental): The eating group will be told specifically to eat a light meal (equivalent to two slices of toasted bread with butter and jam and one cup of coffee or juice) the morning of their surgery, within two hours of their procedure start time.
  Interventions: Other: Non-fasting

INTERVENTIONS:
Other: Non-fasting — Instructing patients to eat before their local-only procedure
  Arms: Not Fasting
Other: Fasting — Instructing patients to fast before their local-only procedure
  Arms: Fasting

SUMMARY:
The purpose of this study is to determine whether eating solid food prior to undergoing a wide awake local-only no tourniquet (WALANT) procedure reduces anxiety in patients or has any effect on outcomes. Patients will be split randomly into two groups and told whether to eat or fast before their procedure. We will then compare levels of anxiety and nausea on the day of the procedure as well as satisfaction with the procedure and other outcome measures at follow-up visits. Our hypothesis is that patients who are instructed to eat before their WALANT procedure will have less anxiety, nausea, and overall higher satisfaction compared to those who are instructed to fast prior to their procedure.

DETAILED DESCRIPTION:
* Patients will initially present for preoperative evaluation in clinic, where they will be approached about whether they are interested in participating. More thorough discussion about risks and benefits will either take place in person at this visit, or over the phone. Consent forms will be signed in person or via Qualtrics/RedCap. If they choose to participate, they will be assigned either to the eating group or the fasting group. Patients in the fasting group will be told to avoid any food past midnight the day before their surgery and any liquids 4 hours before their scheduled surgery. The eating group will be told specifically to eat a light meal (equivalent to two slices of toasted bread with butter and jam, and one cup of coffee or juice) the morning of their surgery, within two hours of their procedure start time. Preoperatively demographic information will be collected via paper forms or via Qualtrics/RedCap both via interview and from medical records, and a pre-operative QuickDASH will be collected as well. All their other preoperative instructions will be consistent with the current protocols.
* On their day of surgery, they will present to the hospital at the pre-arranged time. They will be taken to the preoperative area, where they will be treated in the standard way to prepare them for any procedure. While in the preoperative area, they will be asked whether they ate solid food prior to arrival. They will also be assessed using the Amsterdam Preoperative Anxiety and Information Score and preoperative pain/nausea visual analog score either on paper forms or via Qualtrics/RedCap. Heart rate, blood pressure, and body mass index will also be collected. They will then undergo their procedure the same way regardless of whether they ate.
* Postoperatively, they will be taken to the recovery room. There, they will again be assessed using the Amsterdam Preoperative Anxiety and Information Score and postoperative pain/nausea visual analog score either on paper forms or via Qualtrics/RedCap. Heart rate and blood pressure will also be collected at this time.
* Patients will be followed at regular intervals following their procedure at 2 weeks and 6 weeks. At their first postoperative visit, patients will be assessed using the surgical satisfaction-8 scores either on paper forms or via Qualtrics/RedCap.
* Patients will also be given the Disabilities of the Arm, Shoulder, and Hand (QuickDASH) to complete at their second postoperative visit at approximately 6 weeks either on paper forms or via Qualtrics/RedCap.
* Patient data will be collected until 6 months post operatively. Complications such as wound healing, infections, medication side effects will be included in data collection, these will be collected from medical records only and no further study surveys or interventions will be performed after the second postoperative visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing wide-awake, local anesthetic-only, no-tourniquet (WALANT) procedures with the lead researcher.

Exclusion Criteria:

* Patients with insulin-dependent diabetes or allergy to local anesthesia, < 18 years of age, patients unable to follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Score | Prior to and immediately following the procedure
  Measure of anxiety

SECONDARY OUTCOMES:
Heart rate | Prior to and immediately following the procedure
  Measure of heart rate
Blood pressure | Prior to and immediately following the procedure
  Measure of blood pressure
Hunger scale | Prior to and immediately following the procedure
  Visual analog scale of hunger (0-10, 10 being more hunger)
Thirst scale | Prior to and immediately following the procedure
  Visual analog scale of thirst (0-10, 10 being more thirst)
Nausea scale | Prior to and immediately following the procedure
  Visual analog scale of nausea (0-10, 10 being more nausea)
Pain scale | Prior to and immediately following the procedure
  Visual analog scale of pain (0-10, 10 being more pain)
Surgical Satisfaction - 8 Score | Approximately 2 weeks after the procedure
  Measure of satisfaction with the procedure
QuickDASH Score | Approximately 6 weeks after the procedure
  Measure of functional status of the upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Kaplan, MD, Principal Investigator — UCI School of Medicine
Locations (1):
- UCI Health Manchester Pavilion, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Connors KM, Guerra SM, Koehler SM. Current Evidence Involving WALANT Surgery. J Hand Surg Glob Online. 2022 Mar 1;4(6):452-455. doi: 10.1016/j.jhsg.2022.01.009. eCollection 2022 Nov. PMID 36420465
- [Background] Shou Wai AT, Abdullah S, Ahmad AA, Yong LC, Jabar FA, Ahmad AR. Prospective Evaluation of Pain and Anxiety Levels Between Wide-Awake Local Anesthesia No Tourniquet and General Anesthesia With Tourniquet in Excision of Wrist Ganglions. J Hand Surg Glob Online. 2022 Aug 5;4(6):414-420. doi: 10.1016/j.jhsg.2022.07.002. eCollection 2022 Nov. PMID 36425368
- [Background] Miller MB, Gabel SA, Gluf-Magar LC, Haan PS, Lin JC, Clarkson JHW. Virtual Reality Improves Patient Experience and Anxiety During In-office Carpal Tunnel Release. Plast Reconstr Surg Glob Open. 2022 Jul 13;10(7):e4426. doi: 10.1097/GOX.0000000000004426. eCollection 2022 Jul. PMID 35919690
- [Background] Shahid S, Saghir N, Saghir R, Young-Sing Q, Miranda BH. WALANT: A Discussion of Indications, Impact, and Educational Requirements. Arch Plast Surg. 2022 Jul 30;49(4):531-537. doi: 10.1055/s-0042-1748659. eCollection 2022 Jul. PMID 35919552
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Bopp C, Hofer S, Klein A, Weigand MA, Martin E, Gust R. A liberal preoperative fasting regimen improves patient comfort and satisfaction with anesthesia care in day-stay minor surgery. Minerva Anestesiol. 2011 Jul;77(7):680-6. Epub 2009 Feb 4. PMID 19190563